CLINICAL TRIAL: NCT02921373
Title: A Phase I Study Evaluating the Feasibility of Using Fluorine-19 Cell Sense to Image Human Peripheral Blood Mononuclear Cells In Vivo
Brief Title: Tracking Peripheral Blood Mononuclear Cells With Fluorine MRI
Acronym: TRACK
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Gregory A. Dekaban (Other)
Collaborators: Western University, Canada (Other); Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Gregory A. Dekaban, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: CS-PBMC-2015-001
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Adverse Reaction to Diagnostic Agents and Kits Nos
Keywords: perfluorocarbon imaging; peripheral blood mononuclear cells; cancer immunotherapy; prostate cancer; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prostate Cancer Patients (Experimental): Up to 6 Male prostate cancer patients with metastatic, castration resistant prostate cancer will be enrolled.
  19F Cell Sense-labeled PBMC (3 million cells) will be injected intradermally into the upper thigh of each participant above the inguinal lymph node. MRI will be used to image the administration site.
  Interventions: Biological: 19F Cell Sense-labeled PBMC; Device: MRI
- Healthy Volunteers (Experimental): Up to 6 male or female healthy volunteers will be enrolled.
  19F Cell Sense-labeled PBMC (3 million cells) will be injected intradermally into the upper thigh of each participant above the inguinal lymph node. MRI will be used to image the administration site.
  Interventions: Biological: 19F Cell Sense-labeled PBMC; Device: MRI

INTERVENTIONS:
Biological: 19F Cell Sense-labeled PBMC — Peripheral blood mononuclear cells (PBMC) will be isolated from patient whole blood samples and labeled in a GMP facility with GMP grade 19F Cell Sense imaging agent.
  These cells will be re-administered to the patient prior to imaging.
Device: MRI — Participants will undergo Magnetic Resonance Imaging (MRI) at 1 hour and 24 hours following PBMC administration

SUMMARY:
Cell-based therapies in the form of stem cell-based or immune cell-based therapies are becoming important treatment options that are either approved for clinical use or are showing promise in clinical trials. One of the issues regarding cell-based therapies is that, once the cells are injected into a subject, there is no easy way to track where they go, assess whether adequate numbers of cells arrive at the intended therapeutic target and for how long they persist at a given location. To address this issue non-invasive imaging methods have been developed using magnetic resonance imaging (MRI). When used with an appropriate cell labelling contrast agent, Cellular MRI can track cells non-invasively in vivo. Detection of cells is accomplished with an inert imaging agent containing the MRI sensitive fluorine-19 (19F) nuclei. The objective of this study is to demonstrate that 19F-MRI is safe to use in humans so that it can subsequently be used to track cell-based immunotherapies in future clinical trials. The long term goal is to be able to quantify immune cell migration to secondary lymphoid tissues and potentially to tumors and correlate to therapeutic outcomes.

DETAILED DESCRIPTION:
Background: None of the currently available Good Manufacturing Practices (GMP)-grade MRI cell labelling agents are approved for use in Canada. There is one iron oxide nanoparticle GMP grade preparation that is commercially available but it is not suitable for labelling the immune cell populations the investigators are interested in tracking in vivo. The investigators have, instead, chosen to develop the commercially available, GMP-grade 19F-based perfluorocarbon, known as Cell Sense, for the purpose of tracking immune cell-based vaccine therapies in vivo. This agent has been successful used in a phase I clinical trial in United States and is approved for a second trial current recruiting, under the oversight of the FDA.

The cell tracing agent Cell Sense (CS-1000) is an inert, non-metabolizable tracer. As CS-1000 is taken-up and incorporated into the cell traditional pharmacodynamic and pharmacokinetic analyses in animals and humans are not appropriate, as adsorption and biodistribution will vary with cell type, and therefore have not been done. In vitro studies of toxicity towards various cell types did not yield evidence of adverse effects on various cell functions. Cell Sense also was shown to be non-mutagenic using the Ames and Forward thymidine kinase (TK) assays. Some limited skin irritation was observed when >2,500 fold more Cell Sense than expected to be maximally injected into humans was injected intradermally into rats.

Examples of MRI cell tracking labels include superparamagnetic iron oxide nanoparticles and 19F-containing compounds such as perfluorocarbons. The advantage of using cellular MRI to track cells is that a non-radioactive tracer is used that is suitable for longitudinal studies. MRI offers 3D imaging with exquisite soft tissue contrast. The additional advantage of using 19F over iron-based agents is that 19F is a positive, easily quantifiable contrast cell labelling agent. Furthermore, there is no 19F-background MRI signal in humans whereas MRI involving iron can be confounded by different imaging artifacts and it is a negative contrast agent that is difficult to accurately quantify. The investigators are particularly interested in whether immune cells arrive in secondary lymphoid organs such as lymph nodes.

Study Design:

Open label, dose escalating, single centre, phase I study that will accrue (a) 6 healthy adults and (b) 6 prostate cancer patients.

Three healthy adults and three prostate cancer patients will be enrolled into the first cohort. Whole blood (150 ml) will be obtained by venipuncture. After processing of the blood to obtain peripheral blood mononuclear cells (PBMC), half of the PBMC will be treated with Cell Sense for 8-24 hours. Given the robustness of our data using 5 donors during dry runs, the investigators do not propose to compare labeled vs unlabeled cells as release criteria. However, the investigators will be collecting this data for information and research purposes. Three million (3 x 106) Cell Sense labeled autologous PBMC will be administered intradermally to the cohort 1 subjects. The three healthy adults and the 3 prostate cancer subjects will be tested concurrently.

If no grade 2 or higher adverse events are observed with the 1st cohort, concurrent enrolment will proceed to recruit a second set of 3 healthy adult subjects and the second set of 3 prostate cancer patients. The second cohort of subjects will be subjected to the same design but with an escalation of the dose to 2-3 x 107 Cell Sense-labeled autologous PBMC administered intradermally.

Endpoints:

Primary Endpoints:

Determine the feasibility of using Cell Sense to detect and monitor the migration of PBMC in humans

Secondary Endpoints:

* Confirm and further optimize the 19F Cell Sense detection and Hydrogen- 1 (1H) anatomical imaging parameters for imaging using the 19F/1H dual coil.
* Determine if Cell Sense-labeled PBMC migration to the draining lymph node can be detected.
* Determine if the lymph nodes in the area of interest imaged change in size on the injected side compared to the contralateral side.
* Quantify the number of Cell Sense-labeled PBMC detected.
* Evaluate safety parameters (toxicity) as defined by:
* adverse events.
* serious adverse events.
* changes in laboratory determination and vital sign parameters as assessed by medical history, physical examination and clinical laboratory tests.

The following categories will be used to grade any adverse events:

* Grade 1: does not interfere with daily activity,
* Grade 2: interferes with daily activity, no treatment required, except paracetamol,
* Grade 3: prevents daily activity or requires treatment.
* Grade 4: Life-threatening

NIH and FDA (or CTCAE v 4.0) guidelines will be used to determine the severity of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with confirmed adenocarcinoma of the prostate
* No history of skin hypersensitivities or allergies.
* Normal liver functions as defined by alanine aminotransferase (ALT) (3-36 U/L) and aspirate aminotransferase (AST) levels (10-34 U/L)
* Normal kidney function by monitoring urea (2.5-8.0 ηmol/L) and creatine (70-120 μmol/L [for males]) concentrations.
* Normal complete blood count with differential
* Body Weight between 40 and 110 kg (relates to being able to fit in scanner)
* Body Mass Index < 30 (relates to being able to fit in scanner)
* Negative for (HIV, HTLV1&2, Hep A, B, C, syphilis) infection as determined by approved serological testing.

Exclusion Criteria:

* Contraindication to venipuncture and donation of 100-160 mL of blood
* Active infection (not limited to HIV, HTLV1&2, Hep A, B, C, syphilis)
* Participants are on active chemotherapy (not including castrate hormone therapy), radiation therapy or immunosuppressive therapy (i.e. steroid use, anti-transplant rejection drugs, depleting antibodies)
* Participants who are unable to have an MRI scan (e.g. history of head or eye injury involving metal fragments, implanted electrical device (such as a cardiac pacemaker), conductive implants or devices such as skin patches, body piercing or tattoos containing metallic inks, severe heart disease (including susceptibility to heart rhythm abnormalities), claustrophobia, etc.)
* Participants with known allergies to phenol red, β-lactams and β-lactam derivative
* Participants with known allergies to streptomycin sulfate and gentamicin sulfate
* Participants with unforeseen conditions that are deemed unsafe or inappropriate for the study (e.g. participants who are claustrophobic and cannot undergo an MRI) as per the discretion of the principal investigator.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse effects as assessed by CTCAE v4.0 | 12 months

SECONDARY OUTCOMES:
Number of patients with detectable 19F MRI signal at the site of injection | 1hr post injection
  This process will involve testing if the number of PBMC at the site of injection can be visualized and quantified following injection. Signal produced by labeled cells is linearly related to the number of cells. In vivo quantification has been demonstrated in animal modes, but not in a clinical setting to date.
  If necessary, specific imaging parameters will be adjusted to optimize for clinical anatomical and 19F cell tracking imaging.
Number of patients with detectable 19F MRI signal at local lymph nodes | 24 hours post injection
  PBMC are required to migrate to the lymph node for optimum therapeutic effect. Here the investigators will determine if 19F-MRI contains the necessary imaging sensitivity to detect migration.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Dekaban, PhD, Principal Investigator — Robarts Research Institte - Western Universtiy; Paula J Foster, PhD, Principal Investigator — Robarts Research Institte - Western Universtiy; Sowmya Vuswanathan, PhD, Principal Investigator — University Health Network - University of Toronto; Joseph Chin, MD, Study Chair — London Health Research Institute - Western University; Michael Rieder, MD PhD, Study Chair — Robarts Research Institte - Western University; Gary Brahm, MD, Study Chair — London Health Research Institute; Doreen Matsui, MD, Study Chair — Western University; George Dresser, MD, Study Chair — Western University
Locations (1):
- Robarts Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only group data will be presented